CLINICAL TRIAL: NCT03980704
Title: Preoperative Use of the High Protein ONS vs Immunoenhancing ONS in Gastrointestinal Cancer Patients Undergoing Surgery
Brief Title: Preoperative High Protein vs Immunodiet in Surgical Cancer Patients
Acronym: Preop immuno
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanley Dudrick's Memorial Hospital (Other)
Responsible Party: Principal Investigator, Stanislaw Klek, Head of the Unit, Stanley Dudrick's Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Imm1
Record Dates: First submitted 2019-06-05; First posted 2019-06-10 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: General Surgery; Cancer of Colon
Keywords: immunonutrition; preoperative nutrition
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Protein (Active Comparator): Provision of 400 ml per day of high protein oral nutritional supplements
  Interventions: Drug: resource protein
- Immuno ONS (Experimental): Provision of 400 ml per day of immunostimulating oral nutritional supplements
  Interventions: Drug: IMPACT

INTERVENTIONS:
Drug: IMPACT — Administration of oral immunostimulating oral supplement
  Arms: Immuno ONS
Drug: resource protein — Administration of oral high-protein oral supplement
  Arms: High Protein

SUMMARY:
Immunomodulating nutrition is supposed to reduce the number of complications and the legnth of the hospital stay during the postoperative period in patients after major gastrointestinal surgery. The aim of the study is to assess the clinical effect of immunomodulating oral nutrition in patients undergoing resection for gastrointestinal cancer in the group of well-nourished patients.

DETAILED DESCRIPTION:
Between March 1, 2019, and December 31, 2020, a group of 300 well-nourished patients will be enrolled to the study and randomly assigned two one of two groups: A-high protein oral supplements (ONS) and B- immunomodulating ONS. The study is designed to test the hypothesis that immunonutrition and reduce the incidence of infectious complications after upper gastrointestinal surgery; the secondary objective of the study was to evaluate the effect of nutritional intervention on overall morbidity and mortality rates, and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* resectable GI cancer
* written consent

Exclusion Criteria:

* inoperable GI cancer
* known allergy to the drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Infectious complications | 6 months
  Number and type of infectious complications

SECONDARY OUTCOMES:
Surgical complications | 6 months
  Number and type of surgical complications
Length of stay | 14 days
  Hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw Klek, Study Director — Stanley Dudrick's Memorial Hospital
Locations (1):
- Stanley Dudrick's Memorial Hospital, Skawina, Poland

IPD SHARING:
Plan to Share IPD: No